CLINICAL TRIAL: NCT04681170
Title: Phase III, Single Arm, Open Label, International, Multi Centre Study to Evaluate the Efficacy and Safety of Lomitapide in Paediatric Patients With Homozygous Familial Hypercholesterolaemia (HoFH) on Stable Lipid Lowering Therapy
Brief Title: Efficacy and Safety of Lomitapide in Paediatric Patients With Homozygous Familial Hypercholesterolaemia (HoFH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amryt Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APH-19
Record Dates: First submitted 2020-12-07; First posted 2020-12-23 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-06

CONDITIONS: Homozygous Familial Hypercholesterolaemia (HoFH)
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Age 5-10 years (Other): Lomitapide dosing commenced with 2mg at week 1 for 8 Weeks,then increased to 5mg at Week 8±3 days, 10 mg at Week 12±3 days to the maximum allowable dose of 20 mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  Interventions: Drug: Lomitapide
- Age 11-15 years (Other): Lomitapide dosing commenced with 2mg at week 1 for 4 Weeks, then increased to 5mg at Week 4±3 days, 10 mg at Week 8±3 days, 20mg at Week 12±3 days to the maximum allowable dose of 40mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  Interventions: Drug: Lomitapide
- Age 16 to ≤17 years (Other): Lomitapide dosing commenced with 5mg at week 1 for 4 Weeks, then increased to 10mg at Week 4±3 days, 20 mg at Week 8±3 days, 40mg at Week 12±3 days to the maximum allowable dose of 60mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  Interventions: Drug: Lomitapide

INTERVENTIONS:
Drug: Lomitapide — 2mg,5mg, 10mg and 20mg capsules

SUMMARY:
This is a single arm, open label, multi centre phase III study to evaluate the efficacy and long term safety of lomitapide in paediatric patients with HoFH receiving stable lipid lowering therapy (LLT) (including lipoprotein apheresis (LA), when applicable) comprising of the following phases:

* Screening Period (starting at Week 12, i.e. ≤12 weeks prior to Baseline for up to 6 weeks)
* Stratified Enrolment and Start of Run in Period (starting at minimum at Week 6, i.e., 6 weeks prior to Baseline for a minimum of 6 weeks):
* Efficacy Phase (starting at Baseline, i.e. Day [D] 0 for 24 weeks±3 days
* Safety Phase (starting at Week 24±3 days for 80±1 weeks)

DETAILED DESCRIPTION:
Lomitapide has been approved for use in adult patients with HoFH in the European Union (EU) and European Economic Area (EEA), United States of America (USA), Israel, Argentina, Canada, Colombia, and Japan. This study is designed to determine if lomitapide is effective and can be safely administered to paediatric patients with HoFH. If the efficacy and safety so far observed in adults is confirmed in paediatric patients, the potential exists to significantly lower low-density lipoprotein cholesterol (LDL-C) levels in paediatric patients with HoFH. Furthermore, the lower LDL-C levels may reduce atherosclerosis progression and would be expected to benefit these paediatric patients with HoFH.

A single arm, non comparator design has been selected due to the rarity of the disease and because the evaluation of safety variables such as growth and sexual maturation requires longer term observation than would be feasible in the context of a placebo controlled study.

To mitigate the disadvantages of a single arm design, the study includes a Run in Period of at least 6 weeks during which current lipid lowering therapy (LLT) (including lipoprotein apheresis (LA), when applicable) will be stabilised to establish baseline levels allowing each patient to serve as his/her own control. Patients will also remain on stable LLT (including LA, when applicable) during the Efficacy Phase of the study through Week 24±3 days.

ELIGIBILITY:
Inclusion criteria

* Male and female patients aged 5 to ≤17 years with HoFH as defined by any of the following criteria recommended by the Consensus Panel on Familial Hypercholesterolaemia of the European Atherosclerosis Society (EAS) (Cuchel, Bruckert et al. 2014):

  1. Genetic confirmation of 2 mutant alleles at the LDL receptor (LDLR), apo B, Proprotein convertase subtilisin/kexin type 9 (PCSK9), or LDL receptor adapter protein 1 (LDLRAP1) gene locus OR
  2. An untreated LDL C >500 mg/dL (13 mmol/L) or treated LDL C ≥300 mg/dL (8 mmol/L ) together with either Cutaneous or tendon xanthoma before age 10 years or Untreated LDL C levels consistent with heterozygous FH in both parents
* Baseline LDL C on LLT (maximum concentration [Cmax] immediately prior to LA, if applicable)

  1. >160 mg/dL (4.1 mmol/L, no documented cardiovascular disease [CVD]) or
  2. >130 mg/dL (3.4 mmol/L, established CVD defined as aortic valve disease and/or coronary atherosclerosis)
* Body weight ≥15 kg or body mass index (BMI) and height both >10th percentile according to World Health Organization (WHO) Growth Charts for Boys and Girls 5 to 19 Years of Age
* Patient and/or his/her legal representative has/have been informed, has/have read and understood the patient information/informed consent form, and has/have given written informed assent/consent
* Patient and/or his/her legal representative must be able and willing to follow study procedures and instructions, particularly that

  1. LLT (including LA, when applicable) must be stable for at least 6 weeks prior to Baseline (Run in Period) and remain stable through Week 24±3 days (end of Efficacy Phase)
  2. The patient must be compliant with both the low fat diet supplying <20% of energy (calories) from fat or <30 g fat, whichever is the lesser amount starting at the beginning of the Run in Period and the dietary supplement regimen starting at Week 2 of the Run in Period, both continuing until completion of the study
* Postmenarchal female adolescents must be willing to use an effective form of birth control with failure rates <1% per year (e.g., implant, injectable, combined oral contraceptive, intrauterine contraceptive device, sexual abstinence, vasectomy or vasectomised partner) during participation in the study (and at least 4 weeks thereafter). Patients taking oestrogen based oral contraceptives should be advised about possible loss of effectiveness due to diarrhea and/or vomiting. Additional contraceptive measures should be used for 7 days after resolution of symptoms.
* Patient must be in stable physical and mental health at screening

Exclusion criteria

* Other forms of primary hyperlipoproteinaemia and secondary causes of hypercholesterolaemia (e.g., nephrotic syndrome, hypothyroidism)
* Contraindications for the use of lomitapide according to section 4.3 of the European Medicines Agency (EMA) Summary of Product Characteristics (SmPC), such as hypersensitivity to the active substance or to any of the excipients listed in Section 6.1 of the SmPC, known significant or chronic inflammatory bowel disease or malabsorption
* Moderate (Child Pugh B) or severe hepatic impairment (Child Pugh C), active liver disease and/or abnormal liver function tests at screening (AST or ALT >1.5 x upper limit of normal (ULN) and/or total bilirubin >1.5 x ULN in the absence of Gilbert's syndrome or AP >1.5 x ULN [based on appropriate age and gender normal values])
* Serum CK >2 x ULN
* Chronic renal insufficiency with glomerular filtration rate (GFR) <70 mL/min/1.73 m2 calculated using the Schwartz formula
* Uncontrolled hypertension (defined as mean systolic and/or diastolic blood pressure ≥95% of normal for age and sex) despite medical therapy
* New York Heart Association (NYHA) Class III or IV congestive heart failure
* Precocious/delayed puberty or endocrine disorder affecting growth (e.g., hypothyroidism, premature adrenarche)
* History of drug abuse within the last 3 years or habitual alcohol consumption (defined as >1 ounce [28 g] of liquor or 4 ounce glass [113 g] of wine, or the equivalent, ≥3 times per week)
* Life expectancy predicted to be <5 years
* History of a non skin malignancy (with the exception of cervical cancer in situ) within 3 years prior to enrolment
* Treatment with any Investigational Medicinal Product (IMP) within 6 months or 5 times the terminal half life of the corresponding IMP, whichever is longer, before the screening visit
* Patient is a dependent of the sponsor, of the investigational team or his/her immediate family
* Pregnant or nursing women

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (3):
  - Universtiats-Kinderlinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - University Hospital of Cologne, Cologne
  - University Medical Center Hamburg-Eppendorf, Hamburg
- Chaim Sheba Medical Center, Ramat Gan, Israel
- Italy (2):
  - U.O.C. Clinica Medica 1, Padua, Padua
  - Bambino Gesù Children's Hospital,, Roma
- Saudi Arabia (2):
  - King Abdullah International Medical Research Centre (KAIMRC),, Riyadh
  - King Faisal Specialist Hospital, Riyadh
- Spain (3):
  - Hospital Universitari Sant Joan, Reus, Tarragona,
  - Hospital Abente y Lago, A Coruña
  - Hospital Clinico Universitario of Valencia, Valencia
- E.P.S. Fattouma Bourguiba Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masana L, Zambon A, Schmitt CP, Taylan C, Driemeyer J, Cohen H, Buonuomo PS, Alashwal A, Al-Dubayee M, Kholaif N, Diaz-Diaz JL, Maatouk F, Martinez-Hervas S, Mangal B, Lowe S, Cunningham T. Lomitapide for the treatment of paediatric patients with homozygous familial hypercholesterolaemia (APH-19): results from the efficacy phase of an open-label, multicentre, phase 3 study. Lancet Diabetes Endocrinol. 2024 Dec;12(12):880-889. doi: 10.1016/S2213-8587(24)00233-X. Epub 2024 Oct 16. PMID 39426393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female subjects aged 5 to ≤17 years with HoFH were enrolled in the trial at 12 study centres in various countries (3 in Germany, 1 in Israel, 2 in Italy, 2 in Saudi Arabia, 3 in Spain and 1 in Tunisia).
  The first patient first visit was 14 Dec 2020 and the last patient last visit was 06 Jun 2024.
Pre-assignment Details: Subjects underwent assessments to determine eligibility at the Initial Screening Visit (up to 12 weeks prior to Day 0). A total of 46 subjects were enrolled in this study. Of these, 3 subjects were 'Run in' failures and did not complete the Run in Period.). Therefore, a total of 43 (93.5%) subjects entered the Efficacy Phase at Visit 4.
Groups:
- Age 5-10 Years: Lomitapide dosing commenced with 2mg at week 1 for 8 Weeks, then increased to 5mg Week 8±3 days, 10 mg at Week 12±3 days to the maximum allowable dose of 20mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  Lomitapide: 2mg, 5mg, 10mg and 20mg capsules
- Age 11-17 Years: 11-15 years: Lomitapide dosing commenced with 2mg at week 1 for 4 Weeks, then increased to 5mg Week 4±3 days, 10mg at Week 8±3 days, 20mg at week 12±3 days to the maximum allowable dose of 40mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  16-17 years: Lomitapide dosing commenced with 5mg at week 1 for 4 Weeks, then increased to 10mg Week 4±3 days, 20 mg at Week 8±3 days,40mg at week 12±3 days to the maximum allowable dose of 60mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  Lomitapide: 2mg, 5mg, 10mg and 20mg capsules
Period: Pre-run in
Arm/Group | Age 5-10 Years | Age 11-17 Years
Started | 21 | 25
Completed | 21 | 25
Not Completed | 0 | 0
Period: Stratified Enrolment & run-in
Arm/Group | Age 5-10 Years | Age 11-17 Years
Started | 21 | 25
Completed | 20 | 23
Not Completed | 1 | 2
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Open Label Efficacy Phase
Arm/Group | Age 5-10 Years | Age 11-17 Years
Started | 20 | 23
Completed | 20 | 21
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: Open Label Safety Phase
Arm/Group | Age 5-10 Years | Age 11-17 Years
Started | 20 | 21
Completed | 20 | 19
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — AEs and none compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data shown are for participants who completed the baseline visit.
Groups:
- Age 5-10 Years: Lomitapide dosing commenced with 2mg at week 1 for 8 Weeks, then increased to 5mg Week 8±3 days, 10mg at Week 12±3 days to the maximum allowable dose of 20mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  Lomitapide: 2mg, 5mg, 10mg and 20mg capsules
- Age 11-17 Years: 11-15 years: Lomitapide dosing commenced with 2mg at week 1 for 4 Weeks, then increased to 5mg Week 4±3 days, 10mg at Week 8±3 days, 20mg at week 12±3 days to the maximum allowable dose of 40mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  16-17 years: Lomitapide dosing commenced with 5mg at week 1 for 4 Weeks, then increase to 10mg Week 4±3 days, 20 mg at Week 8±3 days, 40mgs at week 12±3 days to the maximum allowable dose of 60mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  Lomitapide: 2mg, 5mg, 10mg and 20mg capsules
- Total: Total of all reporting groups
Arm/Group | Age 5-10 Years | Age 11-17 Years | Total
Number analyzed (Participants) | 20 | 23 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 23 | 43
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.0 (1.54) | 14.0 (1.97) | 10.7 (3.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 10 | 9 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 23 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 23 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 3 | 10 | 13
  Italy | 5 | 2 | 7
  Israel | 3 | 0 | 3
  Tunisia | 5 | 1 | 6
  Germany | 1 | 6 | 7
  Spain | 3 | 4 | 7
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 15.78 (3.338) | 21.52 (4.840) | 18.85 (5.071)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoint: Percent Change in Low-density Lipoprotein Cholesterol (LDL C) at Week 24 Compared to Baseline
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in low density lipoprotein cholesterol (LDL C) at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 24
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Groups:
- All Age Groups: Patients from all age groups have been evaluated together.
- Age 5-10 Years: Patients aged 5-10 years.
- Age 11-17 Years: Patients aged 11-17 years.
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline | -53.910 (25.8287) | -56.529 (26.5401) | -51.633 (25.5658)
Statistical Analysis 1: Comparison: All Age Groups; This was a single-arm study, no comparative group can be assigned; the comparison made for the primary efficacy endpoint is done only between baseline and Week 24 in paediatric subjects (5 to ≤17 years of age). Analysis was made using the one-sample t-test to test the null hypothesis that the percentage change from Baseline was equal to zero against the alternative hypothesis that the percentage change from Baseline was not equal to zero; Test type: Other; p < 0.0001, t-test, 1 sided; Mean Difference (Net) = -53.910, 95% CI 2-sided [-61.8590 to -45.9612]

2. Secondary Outcome: Efficacy Endpoint: Percent Change From Baseline at Week 24 for Various Lipid Parameters
Description: To evaluate the efficacy of lomitapide, as defined by the percent change of the following lipid parameters at the maximum tolerated dose (MTD):
  * Non-high-density lipoprotein cholesterol (Non-HDL-C)
  * Total cholesterol (TC)
  * Very-low-density lipoprotein cholesterol (VLDL-C)
  * Apolipoprotein B (Apo B)
  * TG (Triglycerides)
Time Frame: Baseline through Week 24
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Non-HDL-C | -54.185 (25.0256) | -56.655 (25.9804) | -52.038 (24.5423)
  TC | -50.176 (24.5397) | -52.883 (25.6260) | -47.822 (23.8756)
  VLDL-C | -49.678 (31.6126) | -53.030 (28.0698) | -46.763 (34.7606)
  Apo B | -53.1 (24.76) | -56.2 (24.45) | -50.4 (25.26)
  TG | -49.28 (31.7290) | -52.292 (27.8956) | -46.674 (35.1359)

3. Secondary Outcome: Efficacy Endpoint: Percent Change From Baseline at Week 24 for Lp(a)
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in Lp(a) at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 24
Population: Patients have been evaluated both, as individual age groups and all together. Note: Lp(a) assessment was inadvertently removed from the central laboratory lipid panel during the laboratory set up phase. However, Lp(a) has also been assessed locally, but in various units (mg/dL, g/L, and nmol/L). Sicne Lp(a) concentrations should not be converted from 'nmol/L' to 'mg/dL', or vice versa, and more subjects had values reported in nmol/L, results are presented for the nmol/l only.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 27 | 14 | 13
Percent change from Baseline | -26.757 (32.5675) | -17.248 (36.4246) | -36.996 (25.3314)

4. Secondary Outcome: Percent Change From Baseline at All Other Time Points Through Week 104 for LDL-C
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in LDL-C at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Week 4: number analyzed (Participants) | 42 | 20 | 22
  Week 4 | -1.962 (20.7168) | -5.936 (10.8438) | 1.651 (26.5109)
  Week 8: number analyzed (Participants) | 36 | 17 | 19
  Week 8 | -6.798 (19.1524) | -2.037 (11.8697) | -11.058 (23.3978)
  Week 12: number analyzed (Participants) | 39 | 19 | 20
  Week 12 | -16.638 (23.1978) | -11.742 (16.1686) | -21.289 (27.9618)
  Week 16: number analyzed (Participants) | 33 | 17 | 16
  Week 16 | -36.458 (17.9894) | -32.971 (14.6467) | -40.163 (20.8120)
  Week 20: number analyzed (Participants) | 40 | 19 | 21
  Week 20 | -50.730 (24.8321) | -49.906 (25.1366) | -51.476 (25.1505)
  Week 24: number analyzed (Participants) | 39 | 18 | 21
  Week 24 | -54.602 (26.4557) | -55.825 (27.9112) | -53.554 (25.7903)
  Week 28: number analyzed (Participants) | 38 | 19 | 19
  Week 28 | -55.518 (28.5714) | -57.929 (29.0704) | -53.108 (28.6469)
  Week 32: number analyzed (Participants) | 37 | 20 | 17
  Week 32 | -52.126 (28.7496) | -55.561 (29.7938) | -48.086 (27.8122)
  Week 36: number analyzed (Participants) | 36 | 18 | 18
  Week 36 | -39.823 (32.6612) | -45.072 (32.4809) | -34.574 (32.9076)
  Week 40: number analyzed (Participants) | 40 | 19 | 21
  Week 40 | -49.427 (29.5830) | -52.511 (27.4375) | -46.637 (31.8088)
  Week 44: number analyzed (Participants) | 40 | 20 | 20
  Week 44 | -44.312 (30.3775) | -53.502 (25.8673) | -35.122 (32.3611)
  Week 48: number analyzed (Participants) | 37 | 17 | 20
  Week 48 | -45.315 (29.6526) | -53.965 (23.2741) | -37.963 (32.9544)
  Week 52: number analyzed (Participants) | 35 | 18 | 23
  Week 52 | -44.583 (32.8128) | -52.956 (25.8671) | -35.718 (37.6118)
  Week 56: number analyzed (Participants) | 39 | 20 | 23
  Week 56 | -45.994 (34.3631) | -57.616 (28.1958) | -33.761 (36.6832)
  Week 68: number analyzed (Participants) | 37 | 17 | 20
  Week 68 | -40.831 (37.3821) | -52.220 (24.9512) | -31.151 (43.6898)
  Week 80: number analyzed (Participants) | 38 | 19 | 19
  Week 80 | -42.319 (34.9400) | -49.410 (28.8677) | -35.227 (39.6221)
  Week 92: number analyzed (Participants) | 38 | 20 | 18
  Week 92 | -37.199 (39.6625) | -41.059 (33.6178) | -32.910 (46.0836)
  Week 104: number analyzed (Participants) | 34 | 17 | 17
  Week 104 | -40.159 (30.5026) | -43.168 (25.4634) | -37.150 (35.3743)

5. Secondary Outcome: Percent Change From Baseline at All Other Time Points Through Week 104 for Non-HDL-C
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in Non-HDL-C at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Week 4: number analyzed (Participants) | 42 | 20 | 22
  Week 4 | -1.765 (21.1682) | -5.950 (10.5881) | 2.039 (27.2319)
  Week 8: number analyzed (Participants) | 36 | 17 | 19
  Week 8 | -6.745 (18.6776) | -1.938 (12.1118) | -11.045 (22.5075)
  Week 12: number analyzed (Participants) | 39 | 19 | 20
  Week 12 | -16.497 (22.9850) | -12.039 (15.5376) | -20.733 (28.0917)
  Week 16: number analyzed (Participants) | 33 | 17 | 16
  Week 16 | -36.610 (17.4339) | -33.214 (14.6890) | -40.218 (19.7812)
  Week 20: number analyzed (Participants) | 40 | 19 | 21
  Week 20 | -50.928 (24.3958) | -50.150 (24.7267) | -51.632 (24.6817)
  Week 24: number analyzed (Participants) | 39 | 18 | 21
  Week 24 | -55.033 (25.4297) | -56.006 (27.3439) | -54.200 (24.3220)
  Week 28: number analyzed (Participants) | 38 | 19 | 19
  Week 28 | -55.984 (27.5559) | -58.201 (28.4121) | -53.768 (27.2620)
  Week 32: number analyzed (Participants) | 38 | 20 | 18
  Week 32 | -52.629 (27.8748) | -55.742 (29.1688) | -49.171 (26.7611)
  Week 36: number analyzed (Participants) | 36 | 18 | 18
  Week 36 | -40.574 (31.4293) | -45.464 (31.6491) | -35.685 (31.3277)
  Week 40: number analyzed (Participants) | 40 | 19 | 21
  Week 40 | -50.013 (28.4878) | -52.837 (26.6409) | -47.458 (30.4850)
  Week 44: number analyzed (Participants) | 40 | 20 | 20
  Week 44 | -44.702 (29.8885) | -53.685 (25.3674) | -35.720 (31.9421)
  Week 48: number analyzed (Participants) | 38 | 18 | 20
  Week 48 | -46.770 (29.3974) | -55.873 (23.6964) | -38.577 (32.1148)
  Week 52: number analyzed (Participants) | 35 | 18 | 17
  Week 52 | -45.222 (31.9577) | -53.190 (25.4004) | -36.785 (36.5745)
  Week 56: number analyzed (Participants) | 39 | 20 | 19
  Week 56 | -46.558 (33.4734) | -57.724 (27.7033) | -34.805 (35.6510)
  Week 68: number analyzed (Participants) | 37 | 17 | 20
  Week 68 | -41.576 (36.0854) | -52.331 (24.4942) | -32.433 (42.0777)
  Week 80: number analyzed (Participants) | 38 | 19 | 19
  Week 80 | -42.388 (34.3439) | -49.605 (28.2105) | -35.171 (38.9712)
  Week 92: number analyzed (Participants) | 38 | 20 | 18
  Week 92 | -37.755 (38.4243) | -41.420 (32.7680) | -33.682 (44.4970)
  Week 104: number analyzed (Participants) | 34 | 17 | 17
  Week 104 | -40.511 (30.1102) | -43.555 (24.5843) | -37.468 (35.2966)

6. Secondary Outcome: Percent Change From Baseline at All Other Time Points Through Week 104 for TC
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in TC at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Week 4: number analyzed (Participants) | 42 | 20 | 22
  Week 4 | -2.057 (19.3772) | -5.487 (10.2352) | 1.062 (24.8373)
  Week 8: number analyzed (Participants) | 37 | 18 | 19
  Week 8 | -6.970 (17.6904) | -3.092 (13.2354) | -10.643 (20.7648)
  Week 12: number analyzed (Participants) | 40 | 20 | 20
  Week 12 | -15.961 (21.4313) | -12.881 (15.4304) | -19.041 (26.1667)
  Week 16: number analyzed (Participants) | 33 | 17 | 16
  Week 16 | -33.976 (15.7159) | -30.986 (14.0719) | -37.154 (17.1693)
  Week 20: number analyzed (Participants) | 41 | 20 | 21
  Week 20 | -48.177 (23.2987) | -48.524 (23.7013) | -47.847 (23.4897)
  Week 24: number analyzed (Participants) | 39 | 18 | 21
  Week 24 | -50.922 (24.9738) | -52.132 (26.9234) | -49.885 (23.7998)
  Week 28: number analyzed (Participants) | 38 | 19 | 19
  Week 28 | -51.998 (26.9668) | -54.806 (27.4139) | -49.190 (26.9564)
  Week 32: number analyzed (Participants) | 38 | 20 | 18
  Week 32 | -48.945 (26.2375) | -52.642 (27.5342) | -44.838 (24.8402)
  Week 36: number analyzed (Participants) | 39 | 20 | 19
  Week 36 | -40.643 (30.5125) | -45.656 (29.7175) | -35.365 (31.2402)
  Week 40: number analyzed (Participants) | 41 | 20 | 21
  Week 40 | -45.402 (27.5358) | -46.997 (27.2264) | -43.882 (28.4123)
  Week 44: number analyzed (Participants) | 40 | 20 | 20
  Week 44 | -41.443 (28.3745) | -50.186 (24.6881) | -32.699 (29.7008)
  Week 48: number analyzed (Participants) | 39 | 19 | 20
  Week 48 | -44.164 (27.6987) | -53.422 (22.4426) | -35.369 (29.8353)
  Week 52: number analyzed (Participants) | 36 | 19 | 17
  Week 52 | -42.764 (30.6617) | -51.169 (24.8422) | -33.371 (34.4186)
  Week 56: number analyzed (Participants) | 39 | 20 | 19
  Week 56 | -43.234 (31.3599) | -54.109 (26.0580) | -31.787 (33.0105)
  Week 68: number analyzed (Participants) | 40 | 20 | 20
  Week 68 | -39.672 (33.2025) | -49.108 (24.7124) | -30.236 (38.2710)
  Week 80: number analyzed (Participants) | 39 | 20 | 19
  Week 80 | -40.291 (31.9119) | -48.031 (26.5964) | -32.143 (35.5890)
  Week 92: number analyzed (Participants) | 38 | 20 | 18
  Week 92 | -34.946 (35.8485) | -38.474 (31.6123) | -31.025 (40.6102)
  Week 104: number analyzed (Participants) | 38 | 19 | 19
  Week 104 | -36.017 (32.2354) | -42.430 (24.0856) | -29.605 (38.3282)

7. Secondary Outcome: Percent Change From Baseline at All Other Time Points Through Week 104 for VLDL-C
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in VLDL-C at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Week 4: number analyzed (Participants) | 42 | 20 | 22
  Week 4 | 9.770 (42.2029) | 1.911 (30.6624) | 16.914 (50.1439)
  Week 8: number analyzed (Participants) | 36 | 17 | 19
  Week 8 | 2.857 (34.5887) | 5.190 (35.0331) | 0.771 (35.0086)
  Week 12: number analyzed (Participants) | 39 | 19 | 20
  Week 12 | -7.405 (48.8428) | -6.638 (54.7493) | -8.133 (43.9360)
  Week 16: number analyzed (Participants) | 33 | 17 | 16
  Week 16 | -34.706 (31.6590) | -36.773 (23.3455) | -32.509 (39.3305)
  Week 20: number analyzed (Participants) | 40 | 19 | 21
  Week 20 | -49.068 (25.6958) | -51.943 (26.4251) | -46.467 (25.3796)
  Week 24: number analyzed (Participants) | 39 | 18 | 21
  Week 24 | -53.050 (27.2118) | -54.447 (27.8824) | -51.853 (27.2551)
  Week 28: number analyzed (Participants) | 38 | 19 | 19
  Week 28 | -55.394 (25.0601) | -58.209 (24.3762) | -52.579 (26.0764)
  Week 32: number analyzed (Participants) | 37 | 20 | 17
  Week 32 | -47.899 (55.7396) | -54.787 (28.1792) | -39.796 (76.9320)
  Week 36: number analyzed (Participants) | 36 | 18 | 18
  Week 36 | -46.596 (25.9994) | -47.963 (24.7584) | -45.230 (27.8348)
  Week 40: number analyzed (Participants) | 40 | 19 | 21
  Week 40 | -51.167 (26.7498) | -55.266 (21.3853) | -47.458 (30.8760)
  Week 44: number analyzed (Participants) | 40 | 20 | 20
  Week 44 | -46.750 (33.3163) | -54.803 (19.0837) | -38.696 (42.1620)
  Week 48: number analyzed (Participants) | 37 | 17 | 20
  Week 48 | -38.148 (50.6100) | -50.109 (35.8714) | -27.981 (59.4366)
  Week 52: number analyzed (Participants) | 35 | 18 | 17
  Week 52 | -49.469 (30.0996) | -55.576 (20.3440) | -43.004 (37.4046)
  Week 56: number analyzed (Participants) | 39 | 20 | 19
  Week 56 | -47.051 (32.7429) | -55.292 (28.1394) | -38.375 (35.6732)
  Week 68: number analyzed (Participants) | 37 | 17 | 20
  Week 68 | -47.832 (30.6844) | -50.902 (21.1040) | -45.223 (37.3270)
  Week 80: number analyzed (Participants) | 38 | 19 | 19
  Week 80 | -36.881 (44.5589) | -46.520 (29.3256) | -27.242 (55.0014)
  Week 92: number analyzed (Participants) | 38 | 20 | 18
  Week 92 | -41.368 (31.7375) | -44.652 (23.2247) | -37.718 (39.5304)
  Week 104: number analyzed (Participants) | 34 | 17 | 17
  Week 104 | -39.055 (40.2422) | -44.612 (26.8209) | -33.498 (50.5480)

8. Secondary Outcome: Percent Change From Baseline at All Other Time Points Through Week 104 for Apo B
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in apo B at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Week 4: number analyzed (Participants) | 42 | 20 | 22
  Week 4 | 0.2 (18.99) | -0.5 (16.45) | 0.9 (21.41)
  Week 8: number analyzed (Participants) | 37 | 18 | 19
  Week 8 | -6.5 (19.25) | -2.4 (16.63) | -10.3 (21.15)
  Week 12: number analyzed (Participants) | 40 | 20 | 20
  Week 12 | -15.5 (21.91) | -10.3 (14.37) | -20.8 (26.84)
  Week 16: number analyzed (Participants) | 33 | 17 | 16
  Week 16 | -36.1 (16.70) | -32.6 (14.52) | -39.7 (18.50)
  Week 20: number analyzed (Participants) | 41 | 20 | 21
  Week 20 | -51.6 (24.21) | -52.1 (24.26) | -51.2 (24.76)
  Week 24: number analyzed (Participants) | 39 | 18 | 21
  Week 24 | -54.0 (25.02) | -55.4 (25.73) | -52.7 (24.96)
  Week 28: number analyzed (Participants) | 38 | 19 | 19
  Week 28 | -56.2 (26.17) | -59.2 (25.77) | -53.2 (26.91)
  Week 32: number analyzed (Participants) | 38 | 20 | 18
  Week 32 | -52.0 (28.64) | -55.7 (27.78) | -47.8 (29.80)
  Week 36: number analyzed (Participants) | 39 | 20 | 19
  Week 36 | -43.9 (30.91) | -47.4 (31.45) | -40.3 (30.74)
  Week 40: number analyzed (Participants) | 41 | 20 | 21
  Week 40 | -48.9 (29.11) | -50.6 (27.92) | -47.3 (30.81)
  Week 44: number analyzed (Participants) | 40 | 20 | 20
  Week 44 | -46.1 (28.75) | -53.5 (25.61) | -38.7 (30.42)
  Week 48: number analyzed (Participants) | 39 | 19 | 20
  Week 48 | -48.6 (29.03) | -56.9 (24.99) | -40.7 (30.97)
  Week 52: number analyzed (Participants) | 36 | 19 | 17
  Week 52 | -47.7 (30.16) | -55.4 (26.77) | -39.1 (32.14)
  Week 56: number analyzed (Participants) | 39 | 20 | 19
  Week 56 | -47.1 (33.06) | -57.7 (28.41) | -35.9 (34.63)
  Week 68: number analyzed (Participants) | 40 | 20 | 20
  Week 68 | -44.8 (33.99) | -53.9 (24.92) | -35.7 (39.71)
  Week 80: number analyzed (Participants) | 39 | 20 | 19
  Week 80 | -47.1 (30.58) | -53.7 (25.96) | -40.0 (34.09)
  Week 92: number analyzed (Participants) | 38 | 20 | 18
  Week 92 | -41.8 (35.12) | -45.5 (28.97) | -37.7 (41.39)
  Week 104: number analyzed (Participants) | 38 | 19 | 19
  Week 104 | -44.6 (30.22) | -51.1 (22.42) | -38.1 (35.85)

9. Secondary Outcome: Percent Change From Baseline at All Other Time Points Through Week 104 for TG
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in TG at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104
Population: Patients from all age groups have been evaluated together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Week 4: number analyzed (Participants) | 42 | 20 | 22
  Week 4 | 9.387 (41.7233) | 1.699 (32.1342) | 16.376 (48.5494)
  Week 8: number analyzed (Participants) | 36 | 17 | 19
  Week 8 | 2.649 (35.3115) | 5.577 (36.3036) | 0.029 (35.1807)
  Week 12: number analyzed (Participants) | 39 | 19 | 20
  Week 12 | -7.258 (49.6990) | -6.133 (56.7548) | -8.327 (43.4273)
  Week 16: number analyzed (Participants) | 33 | 17 | 16
  Week 16 | -34.970 (30.2259) | -37.161 (23.9242) | -32.643 (36.4318)
  Week 20: number analyzed (Participants) | 40 | 19 | 21
  Week 20 | -48.989 (25.8872) | -51.346 (27.1808) | -46.856 (25.1360)
  Week 24: number analyzed (Participants) | 39 | 18 | 21
  Week 24 | -52.878 (26.8475) | -53.866 (27.5741) | -52.031 (26.8624)
  Week 28: number analyzed (Participants) | 38 | 19 | 19
  Week 28 | -55.639 (24.6317) | -57.852 (24.1398) | -53.426 (25.5749)
  Week 32: number analyzed (Participants) | 38 | 20 | 18
  Week 32 | -48.697 (54.0396) | -54.381 (28.4810) | -42.380 (73.2737)
  Week 36: number analyzed (Participants) | 36 | 18 | 18
  Week 36 | -46.823 (25.4762) | -48.286 (23.9243) | -45.361 (27.5563)
  Week 40: number analyzed (Participants) | 40 | 19 | 21
  Week 40 | -51.612 (25.9533) | -55.105 (20.8662) | -48.451 (29.9921)
  Week 44: number analyzed (Participants) | 40 | 20 | 20
  Week 44 | -47.065 (31.7596) | -54.885 (18.5911) | -39.245 (39.9507)
  Week 48: number analyzed (Participants) | 38 | 18 | 20
  Week 48 | -39.769 (48.3307) | -51.803 (35.2601) | -28.939 (56.3536)
  Week 52: number analyzed (Participants) | 35 | 18 | 17
  Week 52 | -49.415 (28.4096) | -55.142 (20.0234) | -43.352 (34.8302)
  Week 56: number analyzed (Participants) | 39 | 20 | 19
  Week 56 | -47.707 (32.0150) | -55.648 (26.7620) | -39.349 (35.5528)
  Week 68: number analyzed (Participants) | 37 | 17 | 20
  Week 68 | -48.471 (30.8061) | -51.253 (21.5583) | -46.107 (37.3356)
  Week 80: number analyzed (Participants) | 38 | 19 | 19
  Week 80 | -38.312 (44.1074) | -47.765 (27.6927) | -28.860 (55.1679)
  Week 92: number analyzed (Participants) | 38 | 20 | 18
  Week 92 | -41.549 (30.2027) | -45.140 (23.5731) | -37.558 (36.5005)
  Week 104: number analyzed (Participants) | 34 | 17 | 17
  Week 104 | -39.739 (39.8597) | -45.352 (25.8574) | -34.126 (50.4118)

10. Secondary Outcome: Percent Change From Baseline at All Other Time Points Through Week 104 for Lipoprotein(a) (Lp(a))
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in Lp(a) at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 28 | 14 | 14
Percent change from Baseline
  Week 4: number analyzed (Participants) | 27 | 14 | 13
  Week 4 | 9.660 (63.5768) | 24.269 (84.1451) | -6.072 (23.8773)
  Week 8: number analyzed (Participants) | 22 | 12 | 10
  Week 8 | 1.508 (46.1156) | 13.870 (54.0530) | -13.327 (30.7067)
  Week 12: number analyzed (Participants) | 25 | 14 | 11
  Week 12 | 0.592 (32.5241) | 13.509 (36.2732) | -15.847 (17.2462)
  Week 16: number analyzed (Participants) | 20 | 12 | 8
  Week 16 | -14.648 (26.3140) | -6.564 (29.3156) | -26.775 (15.7748)
  Week 20: number analyzed (Participants) | 24 | 13 | 11
  Week 20 | -16.602 (47.9856) | -3.961 (58.6273) | -31.540 (26.7998)
  Week 24: number analyzed (Participants) | 22 | 11 | 11
  Week 24 | -28.874 (33.5277) | -15.021 (38.1874) | -42.728 (21.9120)
  Week 28: number analyzed (Participants) | 22 | 13 | 9
  Week 28 | -32.628 (32.4047) | -23.314 (36.5744) | -46.081 (20.1331)
  Week 32: number analyzed (Participants) | 24 | 14 | 10
  Week 32 | -20.594 (50.1160) | -27.534 (46.6328) | -10.877 (55.6561)
  Week 36: number analyzed (Participants) | 21 | 14 | 7
  Week 36 | -25.278 (32.4201) | -21.547 (36.2351) | -32.741 (23.6913)
  Week 40: number analyzed (Participants) | 23 | 14 | 9
  Week 40 | -28.257 (34.6849) | -20.400 (39.7347) | -40.480 (21.6021)
  Week 44: number analyzed (Participants) | 20 | 13 | 7
  Week 44 | -30.124 (34.9943) | -25.915 (38.3512) | -37.940 (28.7510)
  Week 48: number analyzed (Participants) | 20 | 13 | 7
  Week 48 | -17.905 (38.3429) | -8.621 (43.0927) | -35.145 (20.2017)
  Week 52: number analyzed (Participants) | 20 | 13 | 7
  Week 52 | -25.635 (42.3832) | -17.270 (47.3261) | -41.170 (27.8522)
  Week 56: number analyzed (Participants) | 20 | 13 | 7
  Week 56 | -22.366 (34.5809) | -14.691 (33.9040) | -36.621 (33.5132)
  Week 68: number analyzed (Participants) | 20 | 13 | 7
  Week 68 | -20.634 (42.9257) | -9.136 (47.0506) | -41.989 (24.2691)
  Week 80: number analyzed (Participants) | 19 | 13 | 6
  Week 80 | -22.659 (42.2271) | -19.135 (48.3708) | -30.295 (26.4884)
  Week 92: number analyzed (Participants) | 18 | 13 | 5
  Week 92 | -22.235 (41.1508) | -16.468 (44.0841) | -37.229 (31.2661)
  Week 104: number analyzed (Participants) | 18 | 13 | 5
  Week 104 | -29.064 (34.5930) | -24.776 (37.6534) | -40.212 (24.8480)

11. Secondary Outcome: Percent Change in TC/HDL-C Ratio From Baseline at All Other Time Points to Week 104
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in TC/HDL-C ratio at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Week 4: number analyzed (Participants) | 42 | 20 | 22
  Week 4 | 0.108 (27.5756) | -10.581 (14.9489) | 9.825 (32.7827)
  Week 8: number analyzed (Participants) | 36 | 17 | 19
  Week 8 | -5.292 (29.1737) | -7.941 (22.3051) | -2.921 (34.6428)
  Week 12: number analyzed (Participants) | 39 | 19 | 20
  Week 12 | -14.501 (27.7248) | -13.695 (24.7560) | -15.266 (30.9105)
  Week 16: number analyzed (Participants) | 33 | 17 | 16
  Week 16 | -33.384 (25.8765) | -38.768 (21.4831) | -27.664 (29.4691)
  Week 20: number analyzed (Participants) | 40 | 19 | 21
  Week 20 | -45.689 (27.0372) | -51.512 (24.7014) | -40.421 (28.5476)
  Week 24: number analyzed (Participants) | 39 | 18 | 21
  Week 24 | -52.155 (25.1906) | -60.174 (23.4381) | -45.281 (25.1244)
  Week 28: number analyzed (Participants) | 38 | 19 | 19
  Week 28 | -50.986 (31.0715) | -59.358 (27.4688) | -42.614 (32.8937)
  Week 32: number analyzed (Participants) | 38 | 20 | 18
  Week 32 | -48.651 (35.4572) | -55.596 (32.8921) | -40.934 (37.5141)
  Week 36: number analyzed (Participants) | 36 | 18 | 18
  Week 36 | -35.860 (35.4801) | -45.043 (34.3337) | -26.677 (35.1331)
  Week 40: number analyzed (Participants) | 40 | 19 | 21
  Week 40 | -43.976 (36.8573) | -56.120 (26.2125) | -32.988 (41.9967)
  Week 44: number analyzed (Participants) | 40 | 20 | 20
  Week 44 | -40.395 (38.1876) | -54.594 (28.2165) | -26.197 (42.1040)
  Week 48: number analyzed (Participants) | 38 | 18 | 20
  Week 48 | -41.720 (36.2674) | -54.921 (27.6549) | -29.839 (39.5405)
  Week 52: number analyzed (Participants) | 35 | 18 | 17
  Week 52 | -43.496 (38.2302) | -57.568 (26.0987) | -28.596 (43.8568)
  Week 56: number analyzed (Participants) | 39 | 20 | 19
  Week 56 | -39.188 (55.5616) | -57.116 (31.2556) | -20.317 (68.9419)
  Week 68: number analyzed (Participants) | 37 | 17 | 20
  Week 68 | -36.874 (41.9020) | -54.241 (26.5277) | -22.111 (47.2744)
  Week 80: number analyzed (Participants) | 38 | 19 | 19
  Week 80 | -39.189 (37.9268) | -49.165 (33.2083) | -29.213 (40.5453)
  Week 92: number analyzed (Participants) | 38 | 20 | 18
  Week 92 | -37.274 (41.0451) | -47.527 (33.5384) | -25.882 (46.3515)
  Week 104: number analyzed (Participants) | 34 | 17 | 17
  Week 104 | -39.358 (34.3438) | -48.484 (25.6330) | -30.233 (39.9837)

12. Secondary Outcome: Percent Change in HDL-C From Baseline at All Other Time Points to Week 104
Description: To evaluate the efficacy of lomitapide, as defined by the percent change in HDL-C at the maximum tolerated dose (MTD)
Time Frame: Baseline through Week 104 week
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Percent change from Baseline
  Week 4: number analyzed (Participants) | 42 | 20 | 22
  Week 4 | 1.428 (19.6280) | 7.659 (16.3760) | -4.236 (20.9511)
  Week 8: number analyzed (Participants) | 36 | 17 | 19
  Week 8 | 4.482 (26.0635) | 12.855 (29.0476) | -3.010 (21.1047)
  Week 12: number analyzed (Participants) | 39 | 19 | 20
  Week 12 | 4.912 (29.1215) | 8.692 (27.6073) | 1.322 (30.7607)
  Week 16: number analyzed (Participants) | 33 | 17 | 16
  Week 16 | 8.059 (31.4604) | 19.392 (24.6238) | -3.984 (34.1243)
  Week 20: number analyzed (Participants) | 40 | 19 | 21
  Week 20 | 6.186 (33.3664) | 17.873 (30.1872) | -4.387 (33.2219)
  Week 24: number analyzed (Participants) | 39 | 18 | 21
  Week 24 | 11.412 (33.0044) | 24.967 (28.3089) | -0.208 (32.8835)
  Week 28: number analyzed (Participants) | 38 | 19 | 19
  Week 28 | 11.154 (36.3133) | 19.883 (27.9809) | 2.425 (42.0330)
  Week 32: number analyzed (Participants) | 38 | 20 | 18
  Week 32 | 15.137 (33.9304) | 19.607 (31.2092) | 10.171 (36.9795)
  Week 36: number analyzed (Participants) | 36 | 18 | 18
  Week 36 | 8.537 (30.2218) | 14.424 (29.7110) | 2.651 (30.4028)
  Week 40: number analyzed (Participants) | 40 | 19 | 21
  Week 40 | 10.043 (35.0097) | 25.145 (32.0096) | -3.620 (32.4844)
  Week 44: number analyzed (Participants) | 40 | 20 | 20
  Week 44 | 12.765 (33.2136) | 22.486 (34.6933) | 3.044 (29.3561)
  Week 48: number analyzed (Participants) | 38 | 18 | 20
  Week 48 | 13.602 (37.5732) | 25.097 (42.3692) | 3.256 (30.0858)
  Week 52: number analyzed (Participants) | 35 | 18 | 17
  Week 52 | 18.032 (35.1079) | 31.674 (35.7852) | 3.587 (28.7665)
  Week 56: number analyzed (Participants) | 39 | 20 | 19
  Week 56 | 11.528 (29.1750) | 21.636 (31.0975) | 0.887 (23.3045)
  Week 68: number analyzed (Participants) | 37 | 17 | 20
  Week 68 | 9.557 (30.6616) | 21.183 (29.0036) | -0.326 (29.1404)
  Week 80: number analyzed (Participants) | 38 | 19 | 19
  Week 80 | 11.606 (30.8242) | 17.203 (31.1788) | 6.010 (30.2457)
  Week 92: number analyzed (Participants) | 38 | 20 | 18
  Week 92 | 17.320 (33.0024) | 29.691 (32.6733) | 3.574 (28.2358)
  Week 104: number analyzed (Participants) | 34 | 17 | 17
  Week 104 | 16.109 (37.2987) | 26.224 (38.9780) | 5.994 (33.6550)

13. Secondary Outcome: Change in LLT From Week 28 Through Week 104
Description: To evaluate the efficacy of lomitapide, as defined by the change in background lipid lowering therapy
Time Frame: Week 28 through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
  Number of subjects treated with LLT at Week 24:
  * All age groups: 41 patients
  * Age 5-10 Years: 20 patients
  * Age 11-17 Years: 21 patients
Measure: Count of Participants; unit: Participants
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 41 | 20 | 21
Participants
  Reduction due to low LDL-C | 2 | 1 | 1
  Discontinuation due to lomitapide increase | 1 | 1 | 0
  Discontinuation due to other reason | 2 | 1 | 1
  Increase due to high LDL-C | 3 | 3 | 0
  Increase due to other reason | 1 | 1 | 0

14. Secondary Outcome: Change in LA From Week 28 Through Week 104
Description: To evaluate the efficacy of lomitapide, as defined by the change in lipoprotein apheresis
Time Frame: Week 28 through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
  Number of subjects treated with LLT (including LA) at Week 24:
  * All age groups: 17 patients
  * Age 5-10 Years: 6 patients
  * Age 11-17 Years: 11 patients
Measure: Count of Participants; unit: Participants
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 17 | 6 | 11
Participants
  Reduction due to Adverse Event (AE) | 1 | 1 | 0
  Reduction due to low LDL-C | 3 | 1 | 2
  Reduction due to other reason | 4 | 3 | 1
  Discontinuation due to low LDL-C | 1 | 1 | 0
  Discontinuation due to other reason | 1 | 1 | 0

15. Secondary Outcome: Number and Percentage of Patients Achieving European Atherosclerosis Society (EAS) Recommended Target (2013) of LDL-C at Any Timepoint Between Baseline and Week 24
Description: To evaluate the efficacy of lomitapide, as defined by the number and percentage of patients achieving EAS recommended target (2013) of LDL-C
Time Frame: Baseline through Week 24
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Count of Participants; unit: Participants
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Participants
  <135 mg/dL - anytime up to Week 24 | 18 | 7 | 11
  <115 mg/dL - anytime up to Week 24 | 16 | 5 | 11
  <110 mg/dL - anytime up to Week 24 | 14 | 4 | 10

16. Secondary Outcome: Number and Percentage of Patients Achieving EAS Recommended Target (2013) of LDL-C at Any Time in the Study
Description: as for outcome 15
Time Frame: Baseline through Week 104
Population: Patients have been evaluated both, as individual age groups and all together.
Measure: Count of Participants; unit: Participants
Arm/Group | All Age Groups | Age 5-10 Years | Age 11-17 Years
Number analyzed (Participants) | 43 | 20 | 23
Participants
  <135 mg/dL - anytime up to week 104 | 23 | 10 | 13
  <115 mg/dL - anytime up to week 104 | 20 | 7 | 13
  <110 mg/dL - anytime up to week 104 | 19 | 6 | 13

17. Other Pre Specified Outcome: Percent Change of Body Mass Index (BMI)
Description: To evaluate the efficacy of lomitapide, as defined by the percent change of BMI
Time Frame: Baseline through Week 104
Population: Patients from all age groups have been evaluated together.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | All Age Groups
Number analyzed (Participants) | 43
Percent change from Baseline
  Week 4 | -1.06 (3.466)
  Week 8: number analyzed (Participants) | 42
  Week 8 | -1.32 (3.954)
  Week 12: number analyzed (Participants) | 41
  Week 12 | -2.36 (4.768)
  Week 16: number analyzed (Participants) | 40
  Week 16 | -2.96 (5.288)
  Week 20: number analyzed (Participants) | 41
  Week 20 | -4.21 (5.708)
  Week 24: number analyzed (Participants) | 41
  Week 24 | -5.04 (5.997)
  Week 28: number analyzed (Participants) | 41
  Week 28 | -4.13 (6.427)
  Week 32: number analyzed (Participants) | 39
  Week 32 | -3.60 (7.145)
  Week 36: number analyzed (Participants) | 40
  Week 36 | -3.92 (7.949)
  Week 40: number analyzed (Participants) | 40
  Week 40 | -3.78 (8.293)
  Week 44: number analyzed (Participants) | 41
  Week 44 | -3.71 (10.406)
  Week 48: number analyzed (Participants) | 41
  Week 48 | -3.92 (10.420)
  Week 52: number analyzed (Participants) | 39
  Week 52 | -3.21 (10.738)
  Week 56: number analyzed (Participants) | 40
  Week 56 | -2.90 (11.520)
  Week 68: number analyzed (Participants) | 40
  Week 68 | -3.00 (12.103)
  Week 80: number analyzed (Participants) | 39
  Week 80 | -1.90 (12.665)
  Week 92: number analyzed (Participants) | 39
  Week 92 | -1.00 (14.108)
  Week 104: number analyzed (Participants) | 39
  Week 104 | -0.11 (13.718)

18. Other Pre Specified Outcome: Lipid Accumulation in the Liver Over Time Measured by Nuclear Magnetic Resonance (NMR) at Baseline and at Week 24, Week 56 and at Week 104
Description: To evaluate the safety of lomitapide, as defined by lipid accumulation in the liver as measured by nuclear magnetic resonance (NMR)
Time Frame: Baseline through Week 104
Population: All subjects were to undergo NMR imaging unless it was contraindicated or not feasible (e.g., due to the need for sedation or general anaesthesia in very young or anxious subjects). In this case, ultrasound scans were to be used at the discretion of the Investigator.
Measure: Count of Participants; unit: Participants
Groups:
- 5-10 Years: Lomitapide dosing commenced with 2mg at week 1 for 8 Weeks, then increased to 5mg Week 8±3 days, 10 mg at Week 12±3 days to the maximum allowable dose of 20mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values.
  Lomitapide: 2mg, 5mg, 10mg and 20mg capsules
- 11-17 Years: 11-15 years: Lomitapide dosing commenced with 2mg at week 1 for 4 Weeks, then increased to 5mg Week 4±3 days, 10mg at Week 8±3 days, 20mg at week 12±3 days to the maximum allowable dose of 40mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values. 16-17 years: Lomitapide dosing commenced with 5mg at week 1 for 4 Weeks, then increased to 10mg Week 4±3 days, 20 mg at Week 8±3 days,40mg at week 12±3 days to the maximum allowable dose of 60mg by Week 16±3 days or the MTD by Week 20±3 days based upon acceptable safety and tolerability criteria in addition to LDL C values. Lomitapide: 2mg, 5mg, 10mg and 20mg capsules
Arm/Group | 5-10 Years | 11-17 Years
Number analyzed (Participants) | 4 | 19
Participants
  Baseline - ≤10% liver fat: number analyzed (Participants) | 2 | 17
  Baseline - ≤10% liver fat | 2 | 16
  Baseline - >10% and ≤20% liver fat: number analyzed (Participants) | 2 | 17
  Baseline - >10% and ≤20% liver fat | 0 | 1
  Baseline - >20% liver fat: number analyzed (Participants) | 2 | 17
  Baseline - >20% liver fat | 0 | 0
  Week 24 - ≤10% liver fat | 1 | 12
  Week 24 - >10% and ≤20% liver fat | 1 | 2
  Week 24 - >20% liver fat | 0 | 1
  Week 24 - No result | 2 | 4
  Week 56 - ≤10% liver fat: number analyzed (Participants) | 3 | 18
  Week 56 - ≤10% liver fat | 0 | 9
  Week 56 - >10% and ≤20% liver fat: number analyzed (Participants) | 3 | 18
  Week 56 - >10% and ≤20% liver fat | 1 | 4
  Week 56 - >20% liver fat: number analyzed (Participants) | 3 | 18
  Week 56 - >20% liver fat | 0 | 0
  Week 56 - No result: number analyzed (Participants) | 3 | 18
  Week 56 - No result | 2 | 5
  Week 104/EoT - ≤10% liver fat: number analyzed (Participants) | 4 | 15
  Week 104/EoT - ≤10% liver fat | 3 | 11
  Week 104/EoT - >10% and ≤20% liver fat: number analyzed (Participants) | 4 | 15
  Week 104/EoT - >10% and ≤20% liver fat | 1 | 4
  Week 104/EoT - >20% liver fat: number analyzed (Participants) | 4 | 15
  Week 104/EoT - >20% liver fat | 0 | 0

19. Other Pre Specified Outcome: Lipid Accumulation in the Liver Over Time Measured by Ultrasound at Baseline and at Week 24, Week 56 and at Week 104
Description: To evaluate the safety of lomitapide, as defined by lipid accumulation in the liver as measured by ultrasound
Time Frame: Baseline through Week 104
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | 5-10 Years | 11-17 Years
Number analyzed (Participants) | 17 | 2
Participants
  Baseline - ≤10% liver fat | 17 | 2
  Baseline - >10% and ≤20% liver fat | 0 | 0
  Baseline - >20% liver fat | 0 | 0
  Week 24 - ≤10% liver fat: number analyzed (Participants) | 15 | 2
  Week 24 - ≤10% liver fat | 15 | 2
  Week 24 - >10% and ≤20% liver fat: number analyzed (Participants) | 15 | 2
  Week 24 - >10% and ≤20% liver fat | 0 | 0
  Week 24 - >20% liver fat: number analyzed (Participants) | 15 | 2
  Week 24 - >20% liver fat | 0 | 0
  Week 24 - No result: number analyzed (Participants) | 15 | 2
  Week 24 - No result | 0 | 0
  Week 56 - ≤10% liver fat: number analyzed (Participants) | 16 | 2
  Week 56 - ≤10% liver fat | 15 | 2
  Week 56 - >10% and ≤20% liver fat: number analyzed (Participants) | 16 | 2
  Week 56 - >10% and ≤20% liver fat | 1 | 0
  Week 56 - >20% liver fat: number analyzed (Participants) | 16 | 2
  Week 56 - >20% liver fat | 0 | 0
  Week 56 - No result: number analyzed (Participants) | 16 | 2
  Week 56 - No result | 0 | 0
  Week 104/EoT - ≤10% liver fat: number analyzed (Participants) | 15 | 1
  Week 104/EoT - ≤10% liver fat | 15 | 0
  Week 104/EoT - >10% and ≤20% liver fat: number analyzed (Participants) | 15 | 1
  Week 104/EoT - >10% and ≤20% liver fat | 0 | 1
  Week 104/EoT - >20% liver fat: number analyzed (Participants) | 15 | 1
  Week 104/EoT - >20% liver fat | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were monitored throughout the study from the time of informed consent through Week 108.
Description: Safety variables included evaluations of AEs, laboratory test results (including assessment of bone health), vital signs, ECGs, pulmonary function tests, and imaging of the liver. In addition, available standard of care echocardiography results were reviewed.
Arm/Group | Age 5-10 Years | Age 11-17 Years
All-Cause Mortality (participants affected / at risk) | 1/20 | 1/23
Serious Adverse Events (participants affected / at risk) | 4/20 | 7/23
Other Adverse Events (participants affected / at risk) | 19/20 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 5-10 Years (N=20) | Age 11-17 Years (N=23)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Aortic valve disease mixed (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Vascular device occlusion (General disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vascular device infection (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age 5-10 Years (N=20) | Age 11-17 Years (N=23)
Alanine aminotransferase increased (Investigations) | 9 (11) | 8 (17)
Aspartate aminotransferase increased (Investigations) | 7 (10) | 8 (18)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 2 (2)
C-reactive protein increased (Investigations) | 3 (5) | 3 (3)
ECG signs of ventricular hypertrophy (Investigations) | 2 (2) | 3 (3)
Transaminases increased (Investigations) | 4 (6) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 2 (4)
Pyrexia (General disorders) | 10 (17) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (9)
Diarrhoea (Gastrointestinal disorders) | 9 (13) | 13 (31)
Abdominal pain (Gastrointestinal disorders) | 8 (23) | 11 (36)
Vomiting (Gastrointestinal disorders) | 10 (22) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (4) | 3 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (3) | 2 (3)
Xanthoma (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
COVID-19 (Infections and infestations) | 4 (5) | 5 (7)
Nasopharyngitis (Infections and infestations) | 3 (6) | 3 (6)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 4 (5)
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2)
Vitamin E increased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Aortic bruit (Investigations) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase (Investigations) | 1 (1) | 0 (0)
Lipoprotein (a) increased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Ultrasound liver abnormal (Investigations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular device occlusion (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0)
Dyspnoea (General disorders) | 0 (0) | 2 (2)
Pharyngeal erythema (General disorders) | 1 (1) | 0 (0)
Rhinorrhoea (General disorders) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arcus lipoides (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrocalcinosis (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Lp(a) analysis was analysed locally as central analysis was only available from January 2022.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators may use the study data only after prior written consent of Amryt Pharmaceuticals DAC. Amryt will review the proposed publication/disclosure prior to submission for publication, presenting, using for instructional purposes or otherwise disclosing the study results. If Amryt supposes the publication/disclosure to risk its ability to patent any invention related to the study, the publication/disclosure will be modified or delayed to allow Amryt to file a patent application.

DOCUMENTS (3):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT04681170/Prot_000.pdf
  • Statistical Analysis Plan: Main Document (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT04681170/SAP_001.pdf
  • Statistical Analysis Plan: Table, Figure and Listing Shells (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT04681170/SAP_002.pdf